CLINICAL TRIAL: NCT05483907
Title: A Phase 2, Randomized, Double-blind, Placebo-controlled, 24-Week Study to Evaluate the Efficacy, Safety, and Tolerability of BBT-877, as Mono- or add-on Therapy, in Patients With Idiopathic Pulmonary Fibrosis (IPF)
Brief Title: To Evaluate the Efficacy, Safety, and Tolerability of BBT-877 in Patients With IPF
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bridge Biotherapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BBT877-IPF-004
Record Dates: First submitted 2022-07-27; First posted 2022-08-02 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Idiopathic Pulmonary Fibrosis
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis | interventions — ATX inhibitor BBT-877

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- BBT-877 (Experimental): 200 mg twice daily (BID)of BBT-877 in patients with IPF, with or without AF approved background therapies (pirfenidone or nintedanib).
  Interventions: Drug: BBT-877
- Placebo (Placebo Comparator): 200 mg twice daily (BID)of Placebo in patients with IPF, with or without AF approved background therapies (pirfenidone or nintedanib).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BBT-877 — BBT-877 24 weeks + Follow-up 4 weeks
  Arms: BBT-877
Drug: Placebo — Placebo 24 weeks + Follow-up 4 weeks
  Arms: Placebo

SUMMARY:
This is a Phase 2, multicenter, randomized, double-blind, placebo-controlled, study to evaluate the efficacy, safety, and tolerability of 200 mg twice daily (BID) of BBT-877 in patients with IPF, with or without AF approved background therapies (pirfenidone or nintedanib).

ELIGIBILITY:
Inclusion Criteria:

* Male patients who have completed family planning or female patient, aged 40 years or older
* Diagnosis of IPF in accordance with American Thoracic Society/European Respiratory Society/Japanese Respiratory Society/Latin American Thoracic Association guidelines for diagnosis in effect at the time of screening
* Chest high-resolution computed tomography (HRCT) performed according to ATS guidelines within 12 months prior to screening and according to minimum requirements for IPF diagnosis by central review based on HRCT and lung biopsy. If no historical acceptable HRCT is available prior to screening, an HRCT can be performed during screening. In both cases, a central reading of the HRCT has to be done as well as a review of lung biopsy slides, if available and potentially supportive for diagnosis.
* Able to walk at least 150 meters during the 6MWT at screening
* Resting oxygen saturation of ≥89% using a maximum of 6 L/min of supplemental oxygen at sea level, and up to 8 L/min at altitude during screening
* FVC ≥45% predicted of normal
* Ratio of forced expiratory volume in the first second (FEV1) to FVC ≥0.7
* Diffusing capacity for the DLCO corrected for hemoglobin ≥30% predicted of normal
* Absence of IPF improvement in the past year, as determined by the investigator
* Patients receiving either pirfenidone or nintedanib, should be on it for at least 3 months and with a stable dose in the 4 weeks prior to screening, OR taking neither pirfenidone

Exclusion Criteria:

* Unable to perform spirometry as per ATS
* Evidence of IPF exacerbation within 3 months prior to and/or during screening
* Evidence of emphysema extent greater than the extent of fibrosis
* Current smoker (tobacco, e-cigarette)
* History of lung transplant or lung volume reduction surgery
* Current immunosuppressive condition
* Estimated life expectancy of less than 12 months or 30 months in the opinion of the investigator
* Congestive heart failure class III or IV according to New-York Heart Association classification
* Pulmonary hypertension (PH) requiring PH specific therapy
* Unstable cardiovascular, pulmonary or other disease within 6 months prior to screening or during the screening period
* Use of other medications likely to interfere with study assessments
* Any other current or prior medical condition, medical or surgical therapies, or clinical trial participation expected to interfere with the conduct of the study or the evaluation of its results

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2023-04-12 (Actual); Primary Completion 2025-01-26 (Actual); Study Completion 2025-02-23 (Actual)

PRIMARY OUTCOMES:
In patients with IPF by measuring the reduction in forced vital capacity (FVC) in mL decline compared to placebo | After 24 weeks of treatment
  Change from baseline in FVC (in mL).

SECONDARY OUTCOMES:
In patients with IPF by measuring the reduction in forced vital capacity (FVC) % predicted decline compared to placebo | After 24 weeks of treatment
  Change from baseline in FVC (%).
To evaluate the effect of on diffusing capacity of lung for carbon monoxide (DLCO) of BBT-877 compared to placebo | After 24 weeks of treatment
  Change from baseline compared to placebo in DLCO
To evaluate the effect on functional exercise capacity (measured by the 6-Minute Walk Test [6MWT]) of BBT-877 compared to placebo | After 24 weeks of treatment
  Change from baseline in functional exercise capacity as measured by change in 6-minute walk distance assessed by the 6MWT
To assess the change in IPF impacts from the patient perspective after 24 weeks of treatment of BBT-877 compared to placebo | after 24 weeks of treatment
  Change in overall respiratory health as measured by the St. George's Hospital Respiratory Questionnaire (SGRQ) total score from baseline and Change in overall IPF impacts as measured by the L-IPF total score from baseline
To assess the change in IPF symptoms from the patient perspective after 24 weeks of treatment of BBT-877 compared to placebo | after 24 weeks of treatment
  Change in overall IPF symptoms as measured by the L-IPF total score from baseline
To evaluate potential effect of BBT-877 on pharmacokinetics (PK)of each antifibrotic(AF)in patients with IPF | 0, 4, 12, 24 weeks of treatment
  Pre-dose and 4 hr-post dose of plasma concentrations
To evaluate the potential effect of each AF on PK of BBT-877 in patients with IPF | 0, 4, 12, 24 weeks of treatment
  Pre-dose and 4 hr-post dose of plasma concentrations.
To assess the safety of BBT-877 compared to placebo | over 24 weeks
  The investigator will be asked to provide an assessment of the severity of the AE using the following categories:
  Mild: Usually transient and may require only minimal treatment or therapeutic intervention. The event does not generally interfere with usual activities of daily living.
  Moderate: Usually alleviated with additional specific therapeutic intervention. The event interferes with usual activities of daily living, causing discomfort but poses no significant or permanent risk of harm to the patient.
  Severe: Interrupts usual activities of daily living, significantly affects clinical status, or may require intensive therapeutic intervention.

CONTACTS AND LOCATIONS:
Locations (44):
- United States (16):
  - Pulmonary Associates P.A., Phoenix, Arizona
  - Southern Arizona VA Health Care System - NAVREF - PPDS, Tucson, Arizona
  - Keck Medical Center of USC, Los Angeles, California
  - VA Palo Alto Health Care System, Palo Alto, California
  - National Jewish Health Main Campus, Denver, Colorado
  - St. Francis Medical Institute - Clinedge, Clearwater, Florida
  - Renstar Medical Research, Ocala, Florida
  - Central Florida Pulmonary Group PA, Orlando, Florida
  - Augusta University, Augusta, Georgia
  - Northwestern Memorial Hospital, Chicago, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - The Lung Research Center, LLC, Chesterfield, Missouri
  - Hannibal Regional Healthcare System-HRMG-Hannibal, Hannibal, Missouri
  - Medical University of South Carolina, Charleston, South Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Premier Pulmonary Critical Care & Sleep Medicine, Denison, Texas
- Australia (3):
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - Royal Brisbane & Women's Hospital, Herston, Queensland
  - Institute for Respiratory Health, Nedlands, Western Australia
- Israel (8):
  - Meir Medical Center, Kfar Saba, Central District
  - Lady Davis Carmel Medical Center, Haifa, Haifa District
  - Hadassah Medical Center, Jerusalem, Jerusalem
  - Tel Aviv Sourasky Medical Center, Ashkelon, Southern District
  - Sheba Medical Center, Ramat Gan, Tel Aviv
  - Barzilai Medical Center, Petah Tikva
  - Rabin Medical Center, Petah Tikva
  - Kaplan Medical Center, Rehovot
- Poland (2):
  - Centrum Dentystyczno Lekarskie Promedica Joanna Markiewicz, Będzin, Silesian Voivodeship
  - Vitamed Galaj i Cichomski sp.j., Bydgoszcz
- South Korea (15):
  - Soon Chun Hyang University Hospital Seoul, Cheonan, Chungcheongnam-do
  - Samsung Medical Center, Seoul, Gangnam-gu
  - The Catholic University of Korea, Bucheon St. Mary's Hospital, Bucheon-si, Gyeonggi-do
  - CHA Bundang Medical Center, CHA University, Seongnam-si, Gyeonggi-do
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Ajou University Hospital, Suwon, Gyeonggi-do
  - Myongji Hospital, Goyang-si, Gyeonggido
  - Pusan National University Yangsan Hospital, Yangsan, Gyeongsangnam-do
  - Gachon University Gil Medical Center, Namdong, Incheon
  - Korea University Anam Hospital, Seoul, Seongbuk-gu
  - The Catholic University of Korea - Eunpyeong St. Mary's Hospital, Yeongdeungpo-dong, Seoul
  - Asan Medical Center, Seoul, Songpa-gu
  - Inje University Haeundae Paik Hospital, Busan
  - Kyung Hee University Hospital, Seoul
  - Severance Hospital Yonsei University, Seoul

REFERENCES:
- [Derived] Maher T, Song JW, Kramer MR, Lancaster L, Corte TJ, Yun J, Kim K, Cho J, Sather LF, George PM, Devaraj A, Jung JH, Jung S. Phase 2 study design and analysis approach for BBT-877: an autotaxin inhibitor targeting idiopathic pulmonary fibrosis. BMJ Open Respir Res. 2025 May 22;12(1):e003038. doi: 10.1136/bmjresp-2024-003038. PMID 40404183